CLINICAL TRIAL: NCT02863315
Title: The Effects of Anodal Transcutaneous Spinal Direct Current Stimulation on Chronic Neuropathic Pain After Spinal Cord Injury: Pilot Study
Brief Title: The Effects of Anodal tsDCS on Chronic Neuropathic Pain After SCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyung-ik Shin, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1604-007-752 SNUH
Record Dates: First submitted 2016-07-28; First posted 2016-08-11 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Neuropathic Pain; Spinal Cord Injury
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: tsDCS
Who Masked: Participant
Masking Description: tsDCS
Oversight: Data Monitoring Committee: No

ARMS (2):
- tsDCS (Experimental): In the tsDCS group, anodal tsDCS will be applied for 20 minutes.
  Interventions: Device: tsDCS
- sham (Placebo Comparator): In sham tsDCS group, the current of anodal tsDCS will be discontinued after 30 s while the power indicator remained on for 20 minutes.
  Interventions: Device: tsDCS

INTERVENTIONS:
Device: tsDCS — Both groups use the same DC-Stimulator Plus (NeuroConn GmbH, Ilmenaus, Germany).
  In the tsDCS group, anode electrode is placed over tenth thoracic vertebra to target spinal cord with 2mA for 20 min, and the cathode (reference) electrode on the head vertex (in the Cz location according to the 10-20 EEG system)
  In sham tsDCS group, anode electrode is placed over tenth thoracic vertebra to target spinal cord with 2mA for 30s, and the cathode (reference) electrode on the head vertex (in the Cz location according to the 10-20 EEG system). The current was discontinued after 30 s while the power indicator remained on.
  Other Names: DC-Stimulator Plus (NeuroConn GmbH, Ilmenaus, Germany)

SUMMARY:
The purpose of this study is to evaluate the analgesic effect of transcutaneous spinal direct current stimulation (tsDCS) applied on spinal cord in patients with spinal cord injury who have chronic neuropathic pain.

DETAILED DESCRIPTION:
Twenty patients with spinal cord injury and bilateral neuropathic pain received single sessions of both sham and anodal tsDCS (2 mA) over tenth thoracic vertebra for 20 min (reference electrodes on the head vertex). Treatment order was randomly assigned. A evaluator rated the pain using the visual analogue scale for pain, Patient Global Assessment and Present Pain Intensity.

ELIGIBILITY:
Inclusion Criteria:

1. cervical or upper thoracic complete motor spinal cord injury, at least 6 months after SCI, 20<=age<90
2. neuropathic pain (LANSS score >= 12), stable chronic pain for at least the three preceding months but not over 5 years
3. score higher than or equal to 4 cm (0 cm = 'no pain' and 10 cm = 'worst possible pain') on the visual ana- logue scale (VAS) for pain perception at the baseline/start of the treatment
4. refractoriness to drugs for pain relief - such as tricyclic antidepressants, antiepileptic drugs, and/or narcot- ics (pain resistant to at least two of these drugs supplied in ade- quate dosages for 6 months)
5. informed consent

Exclusion Criteria:

1. patients with any clinically significant or unstable medical or progressive neurologic disorder
2. contraindication for electrial stimulation such as pacemaker implant
3. Women of childbearing age or pregnancy
4. significant cognitive deficit
5. Syringomyelia
6. neuropsychiatric comorbidity
7. depressive disorder (as indicated by a score of 10 greater on the Beck Depression Inventory)
8. history of substance abuse
9. skin defect under the electrodes
10. progressive neurological disease or other secondary conditions that could impact neuropathic pain

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) for neuropathic pain | Baseline NRS (average NRS over the preceding 24h), Change from Baseline NRS at 0, 60 and 120 minutes after the start of the stimulation
  On a scale of 0 to 10, with 0 being no pain at all and 10 being the worst pain imaginable

SECONDARY OUTCOMES:
Patient Global Assessment (PGA) | Baseline PGA (average PGA over the preceding 24h), Change from Baseline PGA at 0, 60 and 120 minutes after the start of the stimulation
  One of the most widely used patient reported outcomes (PROs) & PGA reflects the global impact of the disease from the patient's perspective
  1. Markedly improved
  2. Moderately improved
  3. Mildly improved
  4. No change
  5. Mildly worse
  6. Moderately worse
  7. Markedly worse
Present Pain Intensity (PPI) | Baseline PPI (average PPI over the preceding 24h), Change from Baseline PPI at 0, 60 and 120 minutes after the start of the stimulation
  Patient's subjective feeling of the intensity of pain right now
  0: No pain
  1. Mild
  2. Discomforting
  3. Distressing
  4. Excruciating
  5. Horrible

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngernyam N, Jensen MP, Arayawichanon P, Auvichayapat N, Tiamkao S, Janjarasjitt S, Punjaruk W, Amatachaya A, Aree-uea B, Auvichayapat P. The effects of transcranial direct current stimulation in patients with neuropathic pain from spinal cord injury. Clin Neurophysiol. 2015 Feb;126(2):382-90. doi: 10.1016/j.clinph.2014.05.034. Epub 2014 Jun 21. PMID 25027640
- [Background] Cogiamanian F, Vergari M, Schiaffi E, Marceglia S, Ardolino G, Barbieri S, Priori A. Transcutaneous spinal cord direct current stimulation inhibits the lower limb nociceptive flexion reflex in human beings. Pain. 2011 Feb;152(2):370-375. doi: 10.1016/j.pain.2010.10.041. Epub 2010 Dec 14. PMID 21159430
- [Background] Parazzini M, Fiocchi S, Liorni I, Rossi E, Cogiamanian F, Vergari M, Priori A, Ravazzani P. Modeling the current density generated by transcutaneous spinal direct current stimulation (tsDCS). Clin Neurophysiol. 2014 Nov;125(11):2260-2270. doi: 10.1016/j.clinph.2014.02.027. Epub 2014 Apr 3. PMID 24784477
- [Background] Cogiamanian F, Vergari M, Pulecchi F, Marceglia S, Priori A. Effect of spinal transcutaneous direct current stimulation on somatosensory evoked potentials in humans. Clin Neurophysiol. 2008 Nov;119(11):2636-40. doi: 10.1016/j.clinph.2008.07.249. Epub 2008 Sep 10. PMID 18786856